CLINICAL TRIAL: NCT07293247
Title: Involved-Station, Intensity-Modulated Post-Operative Radiation Therapy (I²-PORT) for Resected Non-Small Cell Lung Cancer With Residual Mediastinal Adenopathy After Neoadjuvant Therapy (ypN2)
Brief Title: A Study of Targeted Post-Surgery Radiation Therapy for Non-Small Cell Lung Cancer With Remaining Lymph Node Cancer After Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A082402
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immunotherapy; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (SOC chemotherapy/immunotherapy) (Active Comparator): Patients receive SOC chemotherapy or immunotherapy on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI, FDG-PET, and blood sample collection throughout the study.
  Interventions: Drug: Chemotherapy; Other: Immunotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Fludeoxyglucose F-18; Procedure: Biospecimen Collection
- Arm II (I²-PORT, SOC chemotherapy/immunotherapy) (Experimental): Patients undergo I²-PORT QD Monday through Friday over 15-25 fractions over 5-6 weeks. Starting 1-42 days after completion of I²-PORT, patients receive SOC chemotherapy or immunotherapy on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI, FDG-PET, and blood sample collection throughout the study.
  Interventions: Drug: Chemotherapy; Other: Immunotherapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Fludeoxyglucose F-18; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Chemotherapy — Receive standard of care chemotherapy
Other: Immunotherapy — Receive standard of care immunotherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo I²-PORT
  Other Names: IMRT
  Arms: Arm II (I²-PORT, SOC chemotherapy/immunotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Other: Fludeoxyglucose F-18 — Undergo FDG PET scan
  Other Names: PET Scan
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase II trial compares the effect of intensity-modulated post-operative radiation therapy (I²-PORT) followed by standard of care therapy (chemotherapy or immunotherapy) to standard of care therapy alone in treating patients with non-small cell lung cancer (NSCLC) who have remaining lymph node cancer after surgery. Radiation therapy uses high-energy X-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Intensity-modulated radiation therapy is a type of 3-dimensional radiation therapy that uses computer-generated images to show the size and shape of the tumor. Thin beams of radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Adding I²-PORT radiation therapy to standard therapy may be more effective than standard therapy alone in reducing the risk of cancer returning in those who have undergone surgery for NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether intensity-modulated post-operative radiation therapy (I²-PORT) improves disease-free survival (DFS) of patients with R0 resected ypN2 NSCLC compared to standard of care (SOC).

II. To assess whether I²-PORT does not unacceptably increase (by ≥ 6.5 percentage points) the rate of severe (grade ≥ 3 per Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5) late cardiopulmonary toxicity compared to SOC.

SECONDARY OBJECTIVES:

I. 5-year DFS, 2- and 5-year overall survival (OS). II. Local versus (vs.) regional control, rate of distant metastases. III. Acute and late adverse events (AE) rates of specific cardiac, pulmonary, and other toxicities, per CTCAE version 5.0.

IV. Rates of non-mild, moderate, or severe-very severe symptoms per Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE), particularly terms related to cardiopulmonary toxicities, e.g., pain, shortness of breath, cough, wheezing, and heart palpitations.

V. Subset analyses by single vs. multi-station N2 and by adequacy of surgical nodal evaluation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive SOC chemotherapy or immunotherapy on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI), fludeoxyglucose-positron emission tomography (FDG-PET), and blood sample collection throughout the study.

ARM II: Patients undergo I²-PORT once daily (QD) Monday through Friday over 15-25 fractions over 5-6 weeks, starting 4-12 weeks after surgery. Radiation simulation should be performed within 21 days of starting I²-PORT. Starting 1-42 days after completion of I²-PORT, patients receive SOC chemotherapy or immunotherapy on the study. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI, FDG-PET, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
* Histopathologic diagnosis of NSCLC, may have mixed or multiple histologies but no small cell component
* No known EGFR mutation or ALK rearrangement
* No metastatic disease (M0) per most recent PET/CT and head CT/MRI imaging
* No disease progression per CT chest (including upper abdomen as per standard practice) with intravenous (IV) contrast (unless IV contrast is contraindicated) or FDG-PET performed post-neoadjuvant therapy ≤ 90 days prior to registration, either before or after surgery
* No metastatic disease (M0) per head CT/MRI imaging
* Prior treatment with 2-4 cycles of neoadjuvant systemic therapy with any guideline (National Comprehensive Cancer Network [NCCN]) concordant regimen
* Lobectomy or greater oncologic surgical resection within 8 weeks prior to registration
* Complete (R0) resection showing ypN2 disease
* No prior radiotherapy to the lungs or mediastinum
* No treatment with a VEGF inhibitor ≤ 90 days prior to registration or plan to treat with adjuvant systemic therapy including a VEGF inhibitor
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Platelet count ≥ 50,000/mm^3
* Calculated (Calc.) creatinine clearance ≥ 30 mL/min
* Total bilirubin ≤ 3 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 5 x upper limit of normal (ULN)
* Not pregnant, because this study involves radiation therapy, which has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done ≤ 7 days prior to registration is required
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Cardiac function: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* No idiopathic pulmonary fibrosis requiring anti-fibrotic medication: Patients with idiopathic pulmonary fibrosis or inflammatory/interstitial lung disease compromising pulmonary function or requiring ongoing treatment with nintedanib, pirfenidone, or other anti-fibrotic drug are excluded
* HIV-infected patients on effective anti-retroviral therapy with an undetectable viral load within 6 months are eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2026-03-14 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Time from the date of randomization to the date of earliest disease recurrence/progression or deaths of all causes, assessed up to 5 years
  DFS will be analyzed using the Kaplan-Meier methodology and compared between Arm 2 and Arm 1 using a log-rank test stratified by randomization factors. The median DFS for each treatment group will be estimated, and its 80% and 90% confidence intervals will be calculated using the Kaplan-Meier estimator. Additionally, the 24-month DFS rate for each treatment arm, along with its confidence intervals, will be calculated.
Incidence of late grade ≥ 3 cardiopulmonary toxicities | Between 3 and 24 months after protocol therapy
  Will be assessed according to the Common Terminology Criteria for Adverse Events version 5.0. Will be estimated for each treatment group and the difference between the two treatment groups. The confidence intervals of the rate difference at 80% and 90% significance levels will be estimated using the Miettinen-Nurminen method.

SECONDARY OUTCOMES:
5-year DFS | Time from the date of randomization to the date of earliest disease recurrence/progression or deaths of all causes, assessed up to 5 years
  DFS will be analyzed using the Kaplan-Meier methodology and compared between Arm 2 and Arm 1
2-year overall survival (OS) | Time from the date of randomization to death from all causes, assessed up to 2 years
  Will be analyzed using the Kaplan-Meier methodology and compared between Arm 2 and Arm 1 using a log-rank test stratified by randomization factors. Multivariable Cox models will evaluate the treatment effect on survival time and its interaction with baseline covariates, including stage, pre-treatment, histology, and performance status.
5-year OS | Time from the date of randomization to death from all causes, assessed up to 5 years Symptomatic skeletal event free survival (SSE-FS)
  Will be analyzed using the Kaplan-Meier methodology and compared between Arm 2 and Arm 1 using a log-rank test stratified by randomization factors. Multivariable Cox models will evaluate the treatment effect on survival time and its interaction with baseline covariates, including stage, pre-treatment, histology, and performance status.
Patient-reported symptoms | up to 5 years
  Will be assessed using Patient Reported Outcomes - Common Terminology Criteria for Adverse Events and will be evaluated for between-arm differences in proportions of patients with a maximum post-baseline score greater than 0 using Fisher's exact or chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: David Kozono, MD, Study Chair — Alliance for Clinical Trials in Oncology; Jeremy Brownstein, MD, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: No